CLINICAL TRIAL: NCT02237989
Title: Effects Of Native Collagen Type 2 Treatment In Knee Osteoarthritis : A Randomized Controlled Trial
Brief Title: Effects Of Native Collagen Type 2 Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Onur Armağan, Onur Armagan, Medical Doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: FY2001
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis, native collagen type 2, paracetamol
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracetamol (Active Comparator): The 1st group includes 19 patients given 1500mg/day paracetamol for three months
  Interventions: Drug: paracetamol
- native collagen type 2 + paracetamol (Experimental): The 2nd group consists of 20 patients given 1500mg/day paracetamol and 10mg/day native collagen type 2 for three months
  Interventions: Drug: paracetamol+native collagen type 2

INTERVENTIONS:
Drug: paracetamol — 1500 mg
  Arms: paracetamol
Drug: paracetamol+native collagen type 2 — paracetamol (1500 mg) + native collagen type 2 (10mg)
  Arms: native collagen type 2 + paracetamol

SUMMARY:
The aim of this study was to evaluate symptomatic efficacy of native collagen type 2 on joint pain and function and its effects on urinary biological markers related to cartilage degeneration in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
39 patients diagnosed with knee osteoarthritis were separated into two groups. The 1st group includes 19 patients given 1500mg/day paracetamol, the 2nd group consists of 20 patients given 1500mg/day paracetamol and 10mg/day native collagen type 2 for three months.Pretreatment and posttreatment Visual Analog Scale, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), 20-m walking time and Short Form-36 (SF-36), Coll2-1, Coll2-1NO2 and Fibulin-3 levels in urine were compared.

ELIGIBILITY:
Inclusion Criteria:Patients aged 45-70 years with the diagnosis of primary knee OA according to the American College of Rheumatology (ACR) criteria, Kellgren Lawrence radiological stage II or III and knee pain -

Exclusion Criteria:Patients with intraarticular injections or physical therapy within the last year, a previous lower extremity surgery, oral treatment with glucosamine chondroitin or other natural health products within the last month, serious concomitant systemic diseases, peripheral or central neurological disorder, hypersensitivity to paracetamol or se¬vere cardiac, renal, hepatic, hematologic disease

-

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakilan, Specialist, Study Director — Yerkoy State Hospital

REFERENCES:
- [Derived] Bakilan F, Armagan O, Ozgen M, Tascioglu F, Bolluk O, Alatas O. Effects of Native Type II Collagen Treatment on Knee Osteoarthritis: A Randomized Controlled Trial. Eurasian J Med. 2016 Jun;48(2):95-101. doi: 10.5152/eurasianjmed.2015.15030. PMID 27551171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.84 (6.55) | 57.65 (8.73) | 58.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  Turkey | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: the Change From Baseline in Pain During Walking Visual Analog Scale (VAS Walking)
Description: Post treatment comparison of VAS walking between the groups minimum score is 0, maximum score is 10. The clinic of the patient worses when the score increases.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Number analyzed (Participants) | 19 | 20
score on a scale | 3 [0 to 9] | 3 [0 to 9]

2. Secondary Outcome: the Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score
Description: Post treatment comparison of WOMAC between the groups minimum score is 0, maximum score is 100. The clinic of the patient worses when the score increases.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Number analyzed (Participants) | 19 | 20
units on a scale | 52 [24 to 100] | 44 [24 to 100]

3. Secondary Outcome: the Change From Baseline in 20 Meters Walking Time
Description: Post treatment comparison of 20 meters walking time between the groups When the time increases, clinical of the patient worses
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Number analyzed (Participants) | 19 | 20
seconds | 18.84 (4.79) | 18 (3.49)

4. Secondary Outcome: the Change From Baseline in Short Form 36 / Bodily Pain Subgroup
Description: Post treatment comparison of short form 36-bodily pain between groups minimum score 0 maximum score 100 When the score increases, clinic of patient gets better
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Number analyzed (Participants) | 19 | 20
score | 51 [10 to 100] | 52 [10 to 84]

5. Secondary Outcome: the Change From Baseline in Coll2-1 Levels
Description: Post treatment comparison of Coll2-1 levels between groups
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: microgram/ml
Arm/Group | Paracetamol | Native Collagen Type 2 + Paracetamol
Number analyzed (Participants) | 19 | 20
microgram/ml | 130 [22.4 to 596.13] | 155.25 [26.84 to 558.01]

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Treatment Group: 1500 mg/day acetaminophen and 10 mg/day of native type II collagen
- Control Group: 1500 mg/day acetaminophen
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No